CLINICAL TRIAL: NCT04199442
Title: Assessment of Anxiety Incidence Before Regional Anesthesia Achieving.
Brief Title: Anxiety Assessment Before Regional Anesthesia.
Acronym: Stress RA
Status: Terminated | Type: Observational
Why Stopped: Sanitary crisis du to Covid-19
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Pierre Goffin, Principal Investigator, University of Liege
Other Study IDs: 00011
Record Dates: First submitted 2019-12-09; First posted 2019-12-16 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Anxiety Regional Anesthesia Pre-operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We want to assess the level of anxiety of patients who arrive in the operating room before performing regional anesthesia.

DETAILED DESCRIPTION:
When patients arrive in the operating room, we want to submit them a validated questionnaire (APAIS score and STAI-6 score) to assess their anxiety. After that, the care (anesthesia and surgeries) will take place in a very usual way and similar to our standards of care.

ELIGIBILITY:
Inclusion Criteria:

* patient> 18 years
* surgery performed under general anesthesia or not but preceded by a regional anesthesia.

Exclusion Criteria:

* refusal of the patient
* psychiatric disorders (pathological anxiety, psychosis, depression)
* language barrier
* major drug impregnation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who come to the operating room for surgery under regional anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-01-02 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
APAIS score | Achievement of the score on arrival at the operating area (between 15-30 minutes before to realise the regional anesthesia block). Only one determination of the score is made
  anxiety measurement score
STAI-6 score | Achievement of the score on arrival at the operating area (between 15-30 minutes before to realise the regional anesthesia block). Only one determination of the score is made
  anxiety measurement score

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Goffin, Principal Investigator — MontLegia Hospital, Groupe Santé CHC
Locations (1):
- MontLegia Hospital, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Celik F, Edipoglu IS. Evaluation of preoperative anxiety and fear of anesthesia using APAIS score. Eur J Med Res. 2018 Sep 11;23(1):41. doi: 10.1186/s40001-018-0339-4. PMID 30205837
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159